CLINICAL TRIAL: NCT06009029
Title: A Multicenter, Single-arm, Prospective Study of SBRT Combined With Zimberelimab (GLS-010) in Patients With Locally Advanced Pancreatic Cancer (SPARK-1 Study)
Brief Title: SBRT Combined With Zimberelimab (GLS-010) in Locally Advanced Pancreatic Cancer (SPARK-1 Study)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPARK-1
Record Dates: First submitted 2023-08-09; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Locally Advanced Pancreatic Cancer; SBRT; Zimberelimab
MeSH Terms: interventions — Radiosurgery; zimberelimab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT Combined With Zimberelimab (Experimental): Patients diagnosed with locally advanced pancreatic cancer are treated with SBRT combined with Zimberelimab
  Interventions: Radiation: Stereotactic body radiation(SBRT); Drug: Zimberelimab (GLS-010)

INTERVENTIONS:
Radiation: Stereotactic body radiation(SBRT) — SBRT: 7-10 Gy/F, 5 doses
  Zimberelimab: 240mg d1 iv Q21D, within 7 days after SBRT completion. Receiving a minimum of six cycles of treatment, or disease progression or intolerable toxic side effects.
Drug: Zimberelimab (GLS-010) — Zimberelimab (GLS-010),240mg d1 iv Q21D
  Other Names: Immunotherapy

SUMMARY:
This trial is designed to investigate the efficacy and safety of patients with locally advanced pancreatic cancer by SBRT combined with Zimberelimab(GLS-010).

DETAILED DESCRIPTION:
This a prospective, single-arm, multicenter study evaluating the efficacy and safety of stereotactic radiotherapy (SBRT) and Zimberelimab(GLS-010) in patients with pancreatic cancer. The primary endpoint is OS, and the secondary are PFS, ORR,DCR and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old.
* Locally advanced pancreatic cancer confirmed histologically and defined according to the NCCN Pancreatic Cancer Guidelines v1.2022 as unresectable or surgically declined.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* The expected survival ≥ 3 months.
* At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
* Patient must have adequate organ function defined by the study-specified laboratory tests.

Exclusion Criteria:

* Tumor invasion of the gastrointestinal tract, specifically pancreatic tumor or lymph node metastasis invading the gastrointestinal parenchyma.
* Woman who are pregnant or breastfeeding.
* Has a known additional malignancy within the past 5 years, except for cured skin cancer and cervical carcinoma in situ.
* Patients who have received prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
* Contraindications to immunotherapy.
* Other conditions that investigator decides not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival (PFS) will be defined as the elapsed time from the first date of study treatment until death from any cause. For patients who remain alive, follow-up time will be censored at the date of last disease assessment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per RECIST 1.1) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Objective response rate (ORR) | 2 years
  Disease control rate will be defined as PR +CR rate.
Disease Control Rate (DCR) | 2 years
  Disease control rate will be defined as objective response rate + steady disease rate.
Adverse Events | 2 years
  Based on NCI-CTC AE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, M.D., Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No